CLINICAL TRIAL: NCT04506736
Title: Open Lung Approach Versus Conventional Protective Ventilation in Obese Patients Undergoing Open Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Open Lung Approach Versus Conventional Protective Ventilation in Obese Patients Undergoing Open Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 6204
Record Dates: First submitted 2020-07-24; First posted 2020-08-10 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Abdominal Surgery; Obese Patients
Keywords: Open lung approach; conventional ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPV spontanous ventilation (Active Comparator): The patients will be ventilated using volume controlled ventilation (7ml/kg tidal volume) with addition of 5 cm H₂O fixed PEEP till the end of the surgery .
  Interventions: Other: spontanous ventilation
- OLA open lung ventilation (Active Comparator): The patients will undergo ARM followed by personalized PEEP.
  Interventions: Other: ARM

INTERVENTIONS:
Other: ARM — The ARM is performed by setting the peak inspiratory pressure to 45 cmH₂O then changing the mode of ventilation to pressure controlled ventilation (PCV) with the inspiratory pressure set to give a tidal volume equal to that given during VCV, I:E ratio of 1:1 and a PEEP of 5 cmH₂O. The PEEP level is then increased in 5 cmH₂O steps every minute till it reaches 20 cmH₂O and inspiratory pressure is increased to get an airway opening pressure (inspiratory pressure + PEEP) of 40 cmH₂O which is maintained for one minute after which the ventilation returned to the original setting except for the PEEP level which is kept at 20 cmH₂O.
  The titration of individualized PEEP is done by decremental reduction of the 20 cmH₂O PEEP level in 2 cmH₂O steps every 2 minutes and measuring static compliance of the respiratory system (CRS) at each step.
  Other Names: followed by personalized PEEP.
  Arms: OLA open lung ventilation
Other: spontanous ventilation — volume controlled ventilation (7ml/kg tidal volume) with addition of 5 cm H₂O fixed PEEP till the end of the surgery .
  Arms: SPV spontanous ventilation

SUMMARY:
the purpose of this study is to compare open lung approach versus conventional protective ventilation in obese patients undergoing open abdominal surgery

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into 2 groups each one containing 24 patients Group SPV: will be ventilated using volume controlled ventilation (7ml/kg tidal volume) with addition of 5 cm H₂O fixed PEEP till the end of the surgery .

Group OLA: The patients will undergo ARM followed by personalized PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 - 65 years
* BMI between 30-40 kg/m²
* ASA I and II,open elective abdominal surgery which is expected to last for more than 2 hours under general anesthesia and planned to be extubated at the end of surgery

Exclusion Criteria:

* Emergency surgery, pregnancy, chronic obstructive pulmonary disease (FEV1 < 80% of the predicted value)
* active asthma, acute respiratory distress syndrome
* history of pneumothorax, lung cyst, Difficult airway, obstructive sleep apnea,ischemic heart disease, heart failure
* significant arrhythmias and intracranial hypertension. Exposure to radiotherapy and chemotherapy within 2 months before surgery. Advanced Cardiovascular ,liver, renal diseases ischemic heart disease, heart failure, significant arrhythmias and intracranial hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
post-operative pulmonary complications | one week postoperative
  Pulmonary function tests will be done before surgery as a baseline then repeated after the surgery when the patient is fully awake using bedside spirometer in the sitting position.

SECONDARY OUTCOMES:
heart rate | Baseline (before surgery) and intraoperative
  hemodynamic changes
airway pressure | intraoperative
  During mechanical ventilation airway pressures will be continuously monitored.
pulmonary complications. | one week postoperative
  1. Postoperative pulmonary complications which are defined as having one or more of the following: 1.Pneumonia 2. Respiratory failure requiring mechanical ventilation (Postoperative PaO2 < 60 mm Hg on room air, a PaO2:FiO2 ratio < 300 mm Hg) or peripheral oxygen saturation (SpO₂) <90% and requiring oxygen therapy ). 3. Atelectasis requiring bronchoscopic intervention 4. Pulmonary edema ( postoperative acute lung injury or ARDS). 5. Delayed tracheal extubation ( >24 hours postoperatively) or need for reintubation (because of respiratory distress, hypoxia, hypercarbia, or respiratory acidosis). 6. Pneumothorax 7. Bronchospasm (Newly detected refractory expiratory wheeze requiring bronchodilators
length of hospital stay, | postoperative up to one month
  the length of hospital stay, and 30 days mortality.
mean arterial blood pressure | Baseline (before surgery) and intraoperative
  hemodynamic changes
ETCO2 | Baseline (before surgery) and intraoperative
  hemodynamic changes
tidal volume | intraoperative
  During mechanical ventilation tidal volume will be continuously monitored.
SpO2 | Baseline (before surgery) and intraoperative
  hemodynamic changes

CONTACTS AND LOCATIONS:
Overall Officials: Howida A kamal, M.D, Study Director — zagazig U
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Zagazig, Elsharkia,egypt, Egypt